CLINICAL TRIAL: NCT01837082
Title: Randomized, Double-blind, Placebo-controlled Trial of Ferric Carboxymaltose Versus Placebo in Patients With Congestive Heart Failure
Brief Title: Iron in Congestive Heart Failure
Acronym: iCHF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University of Ulm (Other)
Collaborators: RWTH Aachen University (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Mahir Karakas, Dr. med., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iCHF_D.3874; 2012-001134-33 (EudraCT Number)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure; Iron Deficiency; Anemia
Keywords: Heart Failure; Iron Deficiency; Anemia; Ferric Carboxymaltose
MeSH Terms: conditions — Heart Failure; Iron Deficiencies; Anemia | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron (Active Comparator): ferric carboxymaltose
  Interventions: Drug: ferric carboxymaltose
- Placebo (Placebo Comparator): Sodium chloride 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ferric carboxymaltose
  Other Names: Ferinject
  Arms: Iron
Drug: Placebo
  Other Names: Sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
The hypothesis to be tested is whether treatment with intravenous iron (ferric carboxymaltose) will improve left-ventricular ejection fraction in patients with heart failure and iron deficiency as determined by cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure
* At least 18 years of age
* Iron deficiency
* Dyspnea class II or III according to New York Heart Association
* Left-ventricular ejection fraction ≤ 45%

Exclusion Criteria:

* Known sensitivity to any of the products to be administered during dosing
* Immediate need of transfusion
* Patients presenting with an active infection
* Thalassaemia
* Other forms of microcytic anemia not caused by iron deficiency
* History of acquired iron overload
* Need for revascularization, ST-segment elevation myocardial infarction or Non-ST-segment elevation myocardial infarction during the past 3 months (at time of randomization)
* Women who are pregnant or of childbearing age and not using medically acceptable effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the change from baseline to week 12 in left-ventricular ejection fraction as determined by cardiac magnetic resonance imaging. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karakas, MD, Principal Investigator — University of Ulm
Locations (3):
- Germany (3):
  - University of Aachen, Aachen
  - University Heart Center Hamburg, Hamburg
  - University of Ulm, Ulm